CLINICAL TRIAL: NCT02818296
Title: Computerized Cognitive Bias Intervention for Intolerance of Uncertainty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Oglesby01
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Intolerance of Uncertainty; Anxiety
Keywords: Intolerance of uncertainty; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active IU CBM-I (Experimental): This paradigm was designed to train individuals to endorse benign interpretations of ambiguous information and reject negative/threatening interpretations of ambiguous information. Participant's baseline interpretation bias was measured at baseline. Participants then underwent two training phases in which their responses were either reinforced (i.e., they were told they were correct) or punished (i.e., they were told that they were incorrect). Interpretation bias was measured again at post-training.
  Interventions: Behavioral: Active IU CBM-I
- Control CBM-I (Sham Comparator): This paradigm was identical to the active condition except that the word/sentence pairings used were not relevant to IU and/or anxiety.
  Interventions: Behavioral: Control CBM-I

INTERVENTIONS:
Behavioral: Active IU CBM-I
  Arms: Active IU CBM-I
Behavioral: Control CBM-I
  Arms: Control CBM-I

SUMMARY:
This investigation examines the efficacy of a brief, one-session computerized interpretation bias modification paradigm (CBM-I) in the reduction of intolerance of uncertainty. Intolerance of uncertainty is a risk factor for the development and maintenance of various forms of psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Elevated IU interpretation bias at pre-intervention.

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Intolerance of Uncertainty Scale-Short Form | Post-Intervention (directly following the intervention during their baseline appointment) to Month 1 Follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States